CLINICAL TRIAL: NCT07310264
Title: A Phase I, Randomized, Single Ascending Dose, Multiple Ascending Dose, Double-Blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AX-5006 (Aka VT-5006) in Healthy Participants and Participants With Parkinson's Disease.
Brief Title: Research Into the Safety of a New Agent (VT-5006) in People With and Without Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vertero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXL-5006-101; 2025-523254-14-00 (EU CTIS Number); VT-5006-101 (Other: Vertero Therapeutics)
Record Dates: First submitted 2025-11-17; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers (HV); Parkinson's Disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A SAD Active (Experimental): Single Ascending Doses of VT-5006
  Interventions: Drug: VT-5006
- Part A SAD Placebo (Placebo Comparator): Matched Placebo
  Interventions: Drug: Placebo
- Part B MAD Active (Experimental): Multiple ascending doses of VT-5006
  Interventions: Drug: VT-5006
- Part B MAD Placebo (Placebo Comparator): Matched Placebo
  Interventions: Drug: Placebo
- Part C Active Low Dose (Experimental): Low dose VT-5006
  Interventions: Drug: VT-5006
- Part C Active High Dose (Experimental): High dose VT-5006
  Interventions: Drug: VT-5006
- Part C Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VT-5006 — Oral Capsules, Active
  Other Names: AX-5006
  Arms: Part A SAD Active; Part B MAD Active; Part C Active High Dose; Part C Active Low Dose
Drug: Placebo — Oral Capsules, Matched Placebo
  Arms: Part A SAD Placebo; Part B MAD Placebo; Part C Placebo

SUMMARY:
This is a first-in-human (FIH) study of orally administered VT-5006 (also known as AX-5006) in healthy adult volunteers (HVs) and adult participants with Parkinson's disease (PD). The goal of this clinical trial is to learn if VT-5006 is safe and tolerable in healthy volunteers and in participants with PD. It has three Parts (A, B, and C).

Part A: Healthy volunteers aged 18-54 will attend a screening visit, take a single dose of VT-5006 or matching placebo after an overnight fast, stay in the clinic for three nights, and complete a follow-up visit. One group of participants in Part A will be asked to return to the clinic after approximately two weeks, take a single dose of VT-5006 or matching placebo after consuming a high-fat meal and stay in the clinic for another three nights.

Part B: Healthy volunteers aged 18-54 will attend a screening visit, take one dose of VT-5006 or matching placebo each day for seven days after fasting overnight, stay in the clinic for 10 nights, and complete a follow up visit.

Part C: Participants with PD aged 40-80 will attend a screening visit, take one dose of VT-5006 (high dose), VT-5006 (low dose), or matching placebo each day for 28 days, complete two overnight stays in the clinic, attend three clinic visits, one phone call and a follow up visit.

DETAILED DESCRIPTION:
Part A will consist of five single ascending dose (SAD) cohorts, with 8 participants in each cohort. Participants will be randomized to receive either VT-5006 or placebo in a 6:2 ratio. One cohort of 8 participants will complete an additional clinic stay for the purpose of evaluating food effect (FE).

Part B will consist of two multiple ascending dose (MAD) cohorts, with 10 participants in each cohort. Participants will be randomized to receive either VT-5006 or placebo in an 8:2 ratio.

Part C will consist of a single cohort of approximately 24 participants with PD, randomized to receive either VT-5006 (high dose), VT-5006 (low dose) or placebo over 28 days in a 9:9:6 ratio.

ELIGIBILITY:
Parts A and B enroll healthy volunteers; only key entry criteria for Part C are described below.

Inclusion Criteria:

* Diagnosed with PD confirmed by a neurologist within a maximum of 10 years (based of year of diagnosis) prior to screening
* Has a history of GI motility dysfunction or persistent constipation
* Is able to swallow multiple and large capsules without assistance or difficulty, in the opinion of the investigator
* Participants should be on a stable regimen of any prescribed (expect levodopa/carbidopa, levodopa/benserazide or anticholinergic agents) or over-the-counter medications or supplements for at least 60 days prior to enrolment in the study. Participants should not change the dosage or frequency of these medications or supplements while in the study. If changes to medications or supplements are contemplated during the study, the Investigator should be contacted prior to any change.
* Has suitable venous access for blood sampling

Exclusion Criteria:

* Has a known allergy or hypersensitivity to any component of the formulation of VT-5006 or matching placebo, or history of severe allergy or anaphylaxis to a drug, food, or other exposure
* Participants taking levodopa/carbidopa or levodopa/benserazide must remain on a stable dose and regimen from at least 21 days prior to Day 1 visit to end of study (EOS) visit. Other treatments for PD symptoms may be allowed at the discretion of the medical monitor
* Has any clinically significant arrhythmia(s) on ECG; specifically, the participant's corrected QT interval (QTcf) (Fridericia's correction) is >450 ms for males or >470 ms for females
* Has clinically significant abnormalities, as judged by the investigator, in laboratory test results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis). In the case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility or judged to be clinically irrelevant for healthy participants
* Has any of the following test results: a serum total bilirubin value >1.5 x upper limit of normal (ULN); a serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value 2x ULN. As an exception, participants that present with elevated bilirubin in the absence of elevations in ALT or AST that fits the pattern of Gilbert's syndrome may be enrolled after discussion with the medical monitor if their conjugated bilirubin is not or slightly elevated and the level is considered to be not clinically significant.
* Any history of lumbar surgery for any reason (e.g. herniated disc) that in the opinion of the Investigator would interfere with or pose risks to a lumbar puncture procedure
* Other contraindications to having a lumbar puncture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs) | Part A: Up to 8 days; Part B: Up to 15 days; Part C: Up to 35 days;
  Incidence of treatment-emergent AEs (e.g. clinically significant electrocardiogram, vital signs and physical examination abnormalities; clinically significant changes on the Columbia-Suicide Severity Rating Scale [C-SSRS]).

SECONDARY OUTCOMES:
Plasma pharmacokinetic (PK) parameter: Cmax | Part A: predose, and up to 72 hours postdose; Part B: predose, and up to 37 hours postdose on Days 1 and 7; Part C: predose, and up to 10 hours postdose on Days 1 and 28
  Maximum peak plasma concentration (Cmax)
Plasma PK parameter: Tmax | Part A: predose, and up to 72 hours postdose; Part B: predose, and up to 37 hours postdose on Days 1 and 7; Part C: predose, and up to 10 hours postdose on Days 1 and 28
  Time to Maximum Observed Concentration (Tmax)
Plasma PK parameter: AUClast | Part A: predose, and up to 72 hours postdose; Part B: predose, and up to 37 hours postdose on Days 1 and 7; Part C: predose, and up to 10 hours postdose on Days 1 and 28
  Area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration (AUClast)
Plasma PK parameters: AUCinf | Part A: predose, and up to 72 hours postdose; Part B: predose, and up to 37 hours postdose on Days 1 and 7; Part C: predose, and up to 10 hours postdose on Days 1 and 28
  Area under the concentration-time curve extrapolated to infinity (AUCinf)
Plasma PK parameter: t1/2 | Part A: predose, and up to 72 hours postdose; Part B: predose, and up to 37 hours postdose on Days 1 and 7; Part C: predose, and up to 10 hours postdose on Days 1 and 28
  Terminal-phase elimination half-life (t1/2)
Plasma PK parameter: Apparent CL/F | Part A: predose, and up to 72 hours postdose; Part B: predose, and up to 37 hours postdose on Days 1 and 7; Part C: predose, and up to 10 hours postdose on Days 1 and 28
  Clearance adjusted for bioavailability (CL/F)
Plasma PK parameter: Apparent Vd/F | Part A: predose, and up to 72 hours postdose; Part B: predose, and up to 37 hours postdose on Days 1 and 7; Part C: predose, and up to 10 hours postdose on Days 1 and 28
  Volume of Distribution adjusted for bioavailability (Vd/F)
Food effect on plasma PK: Cmax | Part A: predose and up to 72 hours postdose
  Cmax following a high fat meal
Food effect on plasma PK: Tmax | Part A: predose and up to 72 hours postdose
  Tmax following a high fat meal
Food effect on plasma PK: AUC | Part A: predose and up to 72 hours postdose
  AUC following a high fat meal
Urine PK parameter: CLr | Part A: Up to 72 hours postdose; Part B: Up to 24 hours postdose on Days 1 and 7; Part C: Up to 8 hours postdose on Days 1 and 28
  Renal clearance rate (CLr)
Urine PK parameter: Cumulative Ae(urine) | Part A: Up to 72 hours postdose; Part B: Up to 24 hours postdose on Days 1 and 7; Part C: Up to 8 hours postdose on Days 1 and 28
  Cumulative amount excreted (Ae) in urine
Urine PK parameter: %Cumulative AE | Part A: Up to 72 hours postdose; Part B: Up to 24 hours postdose on Days 1 and 7; Part C: Up to 8 hours postdose on Days 1 and 28
  Percent cumulative amount excreted in urine
Feces PK parameter: Cumulative Ae(feces) | Part A: 0-72 hours postdose; Part B: 0-12 hours and 12-24 hours postdose on Days 1 and 7, and anytime postdose on Day 4; Part C: Anytime postdose on Days 8, 15, 22 and 28
  Cumulative amount excreted (Ae) in feces
Feces PK parameter: %Cumulative AE | Part A: 0-72 hours postdose; Part B: 0-12 hours and 12-24 hours postdose on Days 1 and 7, and anytime postdose on Day 4; Part C: Anytime postdose on Days 8, 15, 22 and 28
  Percent cumulative amount excreted in feces

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No